CLINICAL TRIAL: NCT01734668
Title: Sofia RSV FIA Field Study
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0143-01
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Syncytial Virus
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: In Vitro Diagnostic device to aid in diagnosis

SUMMARY:
The objective of this study is to demonstrate the clinical performance of the Sofia RSV FIA with specimens from symptomatic pediatric subjects who are less than nineteen (19) years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Children less than nineteen (19) years of age can participate (assuming appropriate consent is obtained).
3. Must currently be exhibiting symptoms characteristic of respiratory syncytial virus (RSV) illness.
4. Subjects must present with one or more of the following to be eligible for enrollment:

   * Fever, ≥ 37.8º C (100º F) at present or within past 24 hours
   * Moderate to severe runny nose*
   * Moderate to severe congestion*
   * Decreased appetite
   * Coughing
   * Sneezing*
   * Wheezing
   * Irritability
   * Decreased activity
   * Labored breathing

Exclusion Criteria:

1. Subjects nineteen years of age or older.
2. The parent or legal guardian is unable to understand and consent to participation.
3. Current or prior treatment during this infection with anti-RSV Synagis®.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Recruitment of RSV symptomatic pediatric subjects who are less than nineteen (19) years of age.
Sampling Method: Probability Sample
Enrollment: 2468 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
High level of sensitivity and specificity for performance vs. culture | Culture results within 48 hours of plating
  Clinical performance will be based on comparison of the Sofia RSV FIA results to cell culture.

CONTACTS AND LOCATIONS:
Overall Officials: John D Tamerius, PhD, Study Director — Quidel Corporation
Locations (17):
- United States (17):
  - Best Medical Group, Phoenix, Arizona
  - Santo Nino Medical Clinic, Panorama City, California
  - Genesis Community Health, Boynton Beach, Florida
  - Gentle Medical Associates, Boynton Beach, Florida
  - Pediatrics by the Sea, Delray Beach, Florida
  - Soma Pediatrics, Lake Worth, Florida
  - Adriana Castro, Miami, Florida
  - Lanza Pediatrics, Pensacola, Florida
  - Northeast Pediatrics, St. Petersburg, Florida
  - St. Petersburg Pediatrics, St. Petersburg, Florida
  - Teena Hughes, MD, Tampa, Florida
  - Soma Medical Center, PA Pediatric Site #3, West Palm Beach, Florida
  - Juan E. Batista, MD PA, Pediatric Site #2, West Palm Beach, Florida
  - FastER Urgent Care, Morris Plains, New Jersey
  - Twelve Corners Pediatrics, Rochester, New York
  - Veritas, PA, Belton, Texas
  - Advanced Pediatrics, Vienna, Virginia